CLINICAL TRIAL: NCT06351137
Title: Timecost of Intranasal Versus Intravenous Analgesia in Traumatic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Robert Weenink, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INIV2023
Record Dates: First submitted 2024-03-08; First posted 2024-04-08 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Acute Pain Due to Trauma; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Administration, Intravenous; Administration, Intranasal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV first (Other): Subjects in this group will be instructed to use intravenous administration in the first scenario and use intranasal administration in the second scenario.
  Interventions: Other: Intravenous administration; Other: Intranasal administration
- IN first (Other): Subjects in this group will be instructed to use intranasal administration in the first scenario and use intravenous administration in the second scenario.
  Interventions: Other: Intravenous administration; Other: Intranasal administration

INTERVENTIONS:
Other: Intravenous administration — Analgesia is administered intravenously.
Other: Intranasal administration — Analgesia is administered intranasally using an atomizer.

SUMMARY:
Prehospital treatment of acute traumatic pain is common in military practice. Analgesics are usually administered intravenously (IV). Research from the civil prehospital environment shows that obtaining IV access can be difficult and time consuming, delaying onset of treatment. The challenges for obtaining IV access in the military prehospital setting are even bigger, for example in combat environments. However, this has not been assessed.

Current guidelines also offer alternative routes of administration for analgesics, for example intranasal (IN) administration. IN administration is a fast, easy and effective route of administration. This study determines whether IN administration of analgesia is faster and leads to increased healthcare provider satisfaction compared to IV administration in patients with acute traumatic pain in a simulated military prehospital environment.

ELIGIBILITY:
Inclusion Criteria:

* All navy healthcare personnel attending (simulation) training on prehospital trauma care.

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Time required for administration of analgesic (minutes) | During simulation training (expected <5 minutes)
  Time interval starts when healthcare provider grabs the first required item (e.g. tourniquet, nasal atomizer, ampoule) from the medicine bag. Time interval ends upon completed administration of analgesic.

SECONDARY OUTCOMES:
Total time spent on scene (minutes) | During simulation training (expected <10 minutes)
  Time interval starts when healthcare provider arrives at the patient. Time interval ends when analgesia has been administered and used materials have been disposed.
Time required for obtaining IV access | During simulation training (expected <5 minutes)
  Time interval starts when healthcare provider grabs the first required item (e.g. tourniquet or alcohol wipe) from the medicine bag. Time interval ends when the IV catheter has been taped or flushed (whichever comes last).
Time required preparing IN administration | During simulation training (expected <0.5 minute)
  Time interval starts when healthcare provider grabs the nasal atomizer. Time interval ends when the nasal atomizer has been placed on the syringe.
Satisfaction of the navy nurse regarding the used route of administration. | Directly after completion of simulation training
  This is rated on a 0-10 Likert scale, where 0 represents "extremely unsatisfactory" and 10 represents "extremily satisfactory"

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Hollmann, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No